CLINICAL TRIAL: NCT05586503
Title: EASYII - A Post-Market Clinical Follow-up Study (PMCF) in Patients With Infrarenal Aortic Aneurysm Undergoing Endovascular Stenting With the E-tegra Stent Graft System - Imaging Cohort
Brief Title: EASYII - E-tegra Stent Graft System - Imaging Cohort
Acronym: EASYII
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: JOTEC GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EASYII
Record Dates: First submitted 2022-10-12; First posted 2022-10-19 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Vascular Aneurysm
Keywords: Abdominal; Aorta; Aneurysm; Endovascular; Repair
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ECG-gated CTA (Experimental): For study's purposes, patients will undergo ECG-gated CTA scans instead of CTA scans at pre-operative planning, prior to discharge, 30 days, 6 months, 12 months in order to assess the stent stability and durability as well as the seal of the stent graft during the cardiac cycle and over time. An additional ECG-gated CTA scan may optionally be performed at 24 months if the device fixation and conformability continue up to the 12 months scan.
  Interventions: Diagnostic Test: ECG-gated CTAs

INTERVENTIONS:
Diagnostic Test: ECG-gated CTAs — ECG-gated CTAs will be performed instead of static CTAs comparing to standard of care

SUMMARY:
The objective of the study is to assess the stent stability and durability as well as the seal of the stent graft during the cardiac cycle and over time as well as to evaluate safety and clinical performance of the E-tegra Stent Graft System used in endovascular treatment of infrarenal aortic aneurysm.

DETAILED DESCRIPTION:
In this study, patients will be observed who are treated with an aorto-iliac bifurcated or aorto-uni-iliac configuration of the E-tegra Stent Graft System for the treatment of an infrarenal aortic or aorto-iliac aneurysm. The E-tegra Stent Graft components will be implanted at the discretion of the treating physician according to the local protocols.

EASYII is an interventional, non-randomized, post-market, multicentre study. The EASYII study is conducted to further assess, within the scope of the intended purpose, the E-tegra Stent Graft, including the study specific additional exam (visit at 6 months). The patients will undergo ECG-gated CTA scans instead of static CTA scans at pre-operative planning, prior to discharge, 30 days, 6 months, 12 months in order to assess the stent stability and durability as well as the seal of the stent graft during the cardiac cycle and over time. An additional ECG-gated CTA scan may optionally be performed at 24 months if the stent fixation (barbs) and stent graft conformability continue up to the 12 months scan.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65
* Patient must have an

  * infrarenal aortic aneurysm with diameter ≥ 50 mm in females and ≥ 55 mm in males, or
  * infrarenal aortic aneurysm with 40-50 mm that has increased in size by ≥ 1 cm per year
* Patient is elegible for treatment inside the instructions for use of the E-tegra Stent Graft System
* Patient is able and willing to undergo follow-up imaging and examinations prior to discharge from the hospital, at 30 days and 6 months, 12 months, and annually thereafter until 5 years follow-up
* Patient understands and has signed the Informed Consent Form prior to intervention
* Patient has a life expectancy of at least 5 years

Exclusion Criteria:

* Patient with severe calcification or thrombi in the proximal sealing zone
* Patient with infectious aneurysm
* Patient with inflammatory aneurysm
* Patient with pseudoaneurysm
* Patient with symptomatic aneurysm
* Patient with ruptured or traumatic aneurysm
* Patient with suprarenal, juxtarenal, or pararenal aneurysm
* Patient with aortic dissection
* Patient with a reversed conical neck that is defined as a > 3 mm distal increase over a 15 mm length
* Patient in which the E-tegra Stent Graft System is used in combination with proximal or distal extenders of another company.
* Patient who is planned to be treated with an adjunctive aortic bare metal stent or a fenestrated stent graft
* Patient who is planned to be treated with a chimney / chimneys in the renal or visceral vessels
* Patient who is planned to be treated with an iliac branch device or parallel grafts in the iliac vessels
* Patient with genetic connective tissue disease (e.g. Marfan syndrome or Ehlers-Danlos syndrome)
* Patient with eGFR < 45 ml/min/1.73 m2 before the intervention Patient had or planned to have a major surgical or interventional procedure within 30 days before or 30 days after the planned implantation of the E-tegra Stent Graft System
* Patient with other medical condition that may cause the patient to be non-compliant with the protocol, confound the results, or is associated with a limited life expectancy of less than five years (i.e. heart failure, active malignancy (progressive, stable or partial remission))
* Patient who has been enrolled in another active clinical trial that does not allow inclusion in this trial

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-12-16 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint: | 30 day
  Rate of 30-day mortality
Primary Imaging Endpoint: | 30 day
  Quantifying stent stability and durability as well as the seal of the stent graft during the cardiac cycle and over time at 30 day follow-up

SECONDARY OUTCOMES:
Stent stability and durability as well as the seal of the stent graft during the cardiac cycle based on ECG-gated CT scans | prior to discharge, 6, 12, and optionally at 24 months follow-up
  Stent stability and durability as well as the seal of the stent graft during the cardiac cycle based on ECG-gated CT scans at prior to discharge, 6, 12, and optionally at 24 months follow-up
Stent stability and durability as well as the seal of the stent graft over time based on ECG-gated CT scans | prior to discharge, 6, 12, and optionally at 24 months follow-up
  Stent stability and durability as well as the seal of the stent graft over time based on ECG-gated CT scans at prior to discharge, 6, 12, and optionally at 24 months follow-up
Mortality | 24 hours, 12, 24, 36, 60 months
  Rate of all-cause mortality
Aneurysm-related mortality | 30-day, 12, 24, 36, 60 months
  Rate of aneurysm-related mortality
Aneurysm rupture-related mortality | 30-day, 12, 24, 36, 60 months
  Rate of aneurysm rupture-related mortality
Technical success | 24 hours
  Rate of patients with device technical success
Clinical success | 12 months
  Rate of patients with clinical success
Reintervention | 30-day, 12, 24, 36, 60 months
  Rate of patients with any reintervention
Reintervention-free survival | 12 months
  Rate of patients with reintervention-free survival
Primary limb patency | 30-day, 12, 24, 36, 60 months
  Rate of patients with primary E-tegra Stent Graft limb patency
Secondary limb patency | 30-day, 12, 24, 36, 60 months
  Rate of patients with secondary E-tegra Stent Graft limb patency
Stable aneurysm size | 12, 60 months
  Rate of patients with stable aneurysm size
Decreasing aneurysm size | 12, 60 months
  Rate of patients with decreasing aneurysm size on CTA scan (≤ 5 mm in maximum diameter)
Increasing aneurysm size | 12, 60 months
  Rate of patients with aneurysm growth on CTA scan (≥ 5 mm in maximum diameter)
Major adverse events | 30-day, 12, 24, 36, 60 months
  Rate of patients with major adverse events (aneurysm-related death, aneurysm rupture, new myocardial infarction requiring intervention (percutaneous transluminal coronary angioplasty, bypass), new disabling stroke (mRS ≥ 2), visceral ischemia (bowel ischemia with surgical/endovascular intervention or submission to ICU or bowel necrosis with surgical/endovascular intervention or submission to ICU), new hepatic infarction, new chronic (> 90 days) renal insufficiency/renal failure requiring dialysis, new permanent (> 30 days) paraplegia (modified Tarlov Scale ≤ 2), new permanent (> 30 days) paraparesis (modified Tarlov Scale 3 or 4), lower limb ischemia (increase in Rutherford classification)
Endoleak Type Ia | 12, 60 months
  Rate of patients with Type Ia endoleak
Endoleak Type Ib | 12, 60 months
  Rate of patients with Type Ib endoleak
Endoleak Type II | 12, 60 months
  Rate of patients with Type II endoleak
Endoleak Type III | 12, 60 months
  Rate of patients with Type III endoleak
Endoleak Type IV | 12, 60 months
  Rate of patients with Type IV endoleak
Endoleak of unknown origin | 12, 60 months
  Rate of patients with endoleak of unknown origin
Stent graft migration | 12, 60 months
  Rate of patients with stent graft migration > 10 mm
Dislodgement | 30-day, 12, 24, 36, 60 months
  Rate of patients with stent graft dislodgement (full component separation)
Stent fracture | 12, 60 months
  Rate of patients with stent fracture
Stent graft infection | 30-day, 12, 24, 36, 60 months
  Rate of patients with stent graft infection
Health status | 6, 12, 48 to 60 months
  Rate of patients with the same level of health status as prior to surgery
QoL | 6, 12, 48 to 60 months
  Rate of patients with the same level of QoL as prior to surgery

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Geelkerken, Prof., Principal Investigator — Medisch Spectrum Twente
Locations (4):
- Netherlands (4):
  - Meander Medisch Centrum, Amersfoort
  - Rijnstate Hospital, Arnhem
  - Medisch Spectrum Twente, Enschede
  - Zuyderland Hospital, Heerlen